CLINICAL TRIAL: NCT03287830
Title: Flu2Text: A Multi-Site Study Assessing Text Message Reminders for 2nd Dose of Influenza Vaccine
Brief Title: Flu2Text: Text Message Reminders for 2nd Dose of Influenza Vaccine
Acronym: F2T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); American Academy of Pediatrics (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AAAR4101; R01HD086045-01A1 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-19 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Influenza; Vaccination
Keywords: text message; Short message service (SMS); mHealth
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The care provider, primary statistician and analyst will be blinded to participant status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Text message influenza vaccine reminders
  Interventions: Behavioral: Text message influenza vaccine reminders
- Usual care (No Intervention): Season 2017-18: Usual care has no text message
  Season 2018-19: Usual care includes on text message with a link to American Academy of Pediatrics parenting information page. The purpose is to provide those randomized to usual care with tangible benefit that is not related to the study.

INTERVENTIONS:
Behavioral: Text message influenza vaccine reminders — Text message reminders for second dose of influenza vaccination
  Arms: Intervention

SUMMARY:
This multi-site study assesses the impact of text message reminders on the receipt of the second dose of influenza vaccine, and takes place primarily in practices from the American Academy of Pediatrics (AAP) Pediatric Research in Office Settings (PROS) network.

DETAILED DESCRIPTION:
The study is to be conducted over the 1st season (September 2017-April 2018) as an effectiveness trial and the 2nd (September 2018-April 2019) as a replication study. This approach tests that the intervention effects can be replicated across seasons, during which the severity and incidence of influenza disease may vary. Eligible parents will have a child who received his/her first vaccine dose and is in need of 2 doses that season. Current recommendations require 2 doses for certain children 6 months through 8 years old. Within each practice site, parents will be randomized to receive either: 1) text message reminders embedded with influenza vaccine health-literacy promoting information, or 2) usual care. Randomization is to be stratified by practice site, age (6-23 months, 2-8 years) and language (Spanish, English).

ELIGIBILITY:
Inclusion Criteria:

* Parenting adult (or legal guardian) of a child that:

  * is between 6 months through 8 years at the time of enrollment (or the age for which 2 doses of influenza are recommended should Centers for Disease Control and Prevention (CDC) recommendations change)
  * received 1st dose of influenza vaccine within last 7 days
  * receives care at study site
  * needs 2 doses of influenza vaccine that season as determined by their clinician at the study site
  * plan to continue to receive care through April 30 of that season (to the best of their knowledge) (season 2017-18 only)
* Ability to speak and read English or Spanish
* Has a cell phone that has text message capability

Exclusion Criteria:

* Parenting adult of a child that:

  * already enrolled in the study in this or the previous season
  * will leave practice before end of season (April 30) (to their best knowledge) (2017-18 season only)
* Was told by a health care provider that child should not get the flu shot again due to an allergic reaction or anaphylaxis (2017-18 season only)
* Unable to speak and read English or speak and read Spanish
* Unable to receive or read text messages on their cell phone

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2105 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD, MPH, Principal Investigator — Columbia University; Alex Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - American Academy of Pediatrics, Itasca, Illinois
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Stockwell MS, Shone LP, Nekrasova E, Wynn C, Torres A, Griffith M, Shults J, Unger R, Ware LA, Kolff C, Harris D, Berrigan L, Montague H, Localio AR, Fiks AG. Text Message Reminders for the Second Dose of Influenza Vaccine for Children: An RCT. Pediatrics. 2022 Sep 1;150(3):e2022056967. doi: 10.1542/peds.2022-056967. PMID 35965283

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 1050 | 1055
Completed | 1044 | 1042
Not Completed | 6 | 13
Not completed — Withdrawal by Subject | 1 | 1
Not completed — not meeting inclusion criteria | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 1044 | 1042 | 2086
Age, Customized [Count of Participants; unit: Participants]
  age 6-23 month | 966 | 965 | 1931
  2-8 years | 78 | 77 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 492 | 1013
  Male | 523 | 550 | 1073
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Preferred Language for Texting [Count of Participants; unit: Participants]
  English | 966 | 964 | 1930
  Spanish | 78 | 78 | 156

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Receive Influenza Vaccination by April 30 Each Year
Description: Receipt of second dose influenza vaccine by the end of flu season, which is April 30 each year
Time Frame: Up to receipt of second dose, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 1044 | 1042
Participants | 875 | 843

2. Secondary Outcome: Percentage of Participants Who Receive a Second Vaccination by Day 42 From the Initial Influenza Vaccination
Description: Receipt of second dose influenza vaccine by 42 days after first dose
Time Frame: Up to 42 days after first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 1044 | 1042
Participants | 651 | 580

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/1044 | 0/1042
Serious Adverse Events (participants affected / at risk) | 0/1044 | 0/1042
Other Adverse Events (participants affected / at risk) | 0/1044 | 0/1042

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03287830/Prot_SAP_000.pdf